CLINICAL TRIAL: NCT02072993
Title: A Phase I, Single-center, Single-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral AZD1979 After Single-ascending Doses in Healthy Male Volunteers
Brief Title: A First Time in Man Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1979 in Healthy Males
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopping criteria has been reached
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D3930C00001
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Subjects
Keywords: Phase I, healthy, pharmacokinetics
MeSH Terms: interventions — AZD1979

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1979 (Experimental): Single ascending doses of oral solution AZD1979
  Interventions: Drug: AZD1979
- Placebo (Placebo Comparator): Placebo to match single ascending doses of oral solution AZD1979
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD1979 — Single dose, oral solution administration
  Arms: AZD1979
Drug: Placebo to match — Single dose, oral solution administration
  Arms: Placebo

SUMMARY:
This is a first time in human study to assess the safety and tolerability of AZD1979 following oral administration of single ascending doses in healthy male volunteers. Pharmacokinetics (what the body does to the drug) parameters will also be assessed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male volunteer aged 18 to 50 years
* Have a BMI between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IP
* Any clinically important abnormalities in clinical chemistry, endocrine hormones, hematology, or urinalysis results as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety variables in terms of: Adverse events, clinical laboratory variables, vital signs, electrocardiograms and telemetry, physical examinations, and assessments of anxiety and mood | Up to 62 days

SECONDARY OUTCOMES:
Pharmacokinetics of AZD1979 assessed by means of plasma concentration analyses | up to 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles 6700 W 115th Street, Overland Park, KS USA
Locations (1):
- Research Site, Overland Park, Kansas, United States